CLINICAL TRIAL: NCT05793801
Title: Study of the Impact of Frequency of Changing PICCline Dressings in Patients With Acute Leukemia
Acronym: LEUKA-PICC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIMAO/2021-2/JL-01
Record Dates: First submitted 2023-02-23; First posted 2023-03-31 (Actual); Last update posted 2025-04-14 (Actual); Status verified 2025-04

CONDITIONS: Leukemia
Keywords: Leukemia; Catheters; Dressings
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Intervention Model Description: Prospective two-center randomized open-label controlled pilot study in two parallel groups according to PICCline dressing repair: (i) Control group (every 8 days, see SF2H recommendations), (ii) Experimental group (every 2 days).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): Patients receiving normal management with dressings changed once a week according to the SF2H recommendations.
  Interventions: Other: Dressing change
- Experimental group (Experimental): Patients whose dressings are changed every other day.
  Interventions: Other: Dressing change

INTERVENTIONS:
Other: Dressing change — The patient circuit corresponds to that of usual care.
  Not part of usual patient management:
  * The rhythm of PICCline dressing changes, which differed between the two groups.
  * The collection of pain on a visual analog scale at each dressing change.

SUMMARY:
Peripherally Inserted Central Catheters have been widely used for many years for the administration of chemotherapy to patients with cancer. However, its use entails significant infectious complications and high risks of death.The hypothesis is that increasing the rate of PICCline dressing changes will reduce the occurrence of catheter-related infections.

DETAILED DESCRIPTION:
The PICCline ("Peripherally Inserted Central Catheter") is a central catheter whose brachial insertion is peripheral. It has been widely used for many years for the administration of chemotherapy to patients with cancer. Although its use is growing (2.7 million applications in the USA in 2020), significant infectious complications (especially bacteremia) and even high risks of death are generally associated with it.

In December 2013, the French Society of Hospital Hygiene (SF2H) published a guide of "Recommendations for good practices and management of risks associated with PICC" to help professionals in the use of this device. It states that the rate of dressing repair is set at a maximum of 8 days for a sterile semipermeable transparent dressing; however, this recommendation is based on a questionable level of evidence (grade E level of evidence according to the HAS). In the appendix to this guide, the analysis of the scientific literature does not highlight any articles comparing different dressing repair rates. An observational study was conducted at the University Hospital of Nîmes, in order to determine the rate of infection on PICCline in the Hematology Department. In 2019, out of the 90 PICClines applied (dressing changes every 2 days), 12 infections (local and/or systemic) were noted, i.e. 13.3%.

In order to know the current practices of the different hematology services in France, a survey was conducted to collect protocols for PICCline dressing changes. A total of 23 haematology departments were contacted, 18 of which responded. The observation was made that, although most departments respected the SF2H recommendation (15 out of 18), others proposed different rhythms of care: (a) in the Hematology department at Nîmes University Hospital, dressings are redone every 48 hours, (b) in Montpellier, the frequency was 2 to 3 times a week, (c) in Grenoble, the use of PICCline was abandoned by the medical team who noted too many infections and thromboses associated with this device, and (d) in Toulouse and Strasbourg, the PICCline was used less and less for these same reasons. Moreover, the SF2H recommendations are addressed in a general way to professionals and valid for all patients; but no study can currently affirm that they are applicable to a fragile population of immunocompromised patients in the context of intensive chemotherapy. Hematology patients have a high risk of febrile neutropenia, of around 80%, and this risk of immunosuppression is a non-negligible point in terms of infection prevention during patient management.

In 2019 in France, the Réseau de Prévention des Infections Associées aux Soins launched a campaign to monitor and prevent infections associated with invasive devices. For 3 months, data on the occurrence of infectious episodes were collected in 1001 healthcare facilities. Of the nearly 12,000 bacteremia episodes identified, 25.4% were associated with an intravascular device, 17% of which were PICCline. Moreover, the survey revealed that the highest rates of occurrence were found in the Intensive Care Unit, Oncology and Hematology departments and the prevalence of bacteremia associated with intravascular devices in Hematology represented 39.8%.

Hypothesis : increasing the rate of PICCline dressing changes will reduce the occurrence of catheter-related infections.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of acute myeloblastic leukemia.
* Patient going on intensive induction chemotherapy (causing a "high risk" situation of severe infection defined as profound neutropenia ( Polymorphonuclear neutrophil count <500/mm3) and lasting (>7 days).
* Patients who have had a PICCline placed within the last 24 hours or who require a PICCline placement as part of their hospitalization under optimal hygiene and asepsis conditions.
* Patient housed in a protected environment (flow chamber or Plasmair®).
* Patient who has given free and informed consent.
* Patient affiliated or beneficiary of a health insurance plan.
* Adult patient (≥18 years old).

Exclusion Criteria:

* Patient with PICCline placed during a previous hospitalization.
* Patient in an exclusion period determined by another study.
* Patient under court protection, guardianship or curatorship.
* Patient unable to give consent.
* Patient for whom it is impossible to give informed information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2027-06-06 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of local and/or systemic occurrence of infection on the PICCline in controls | Day 1+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in controls | Day 9+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in controls | Day 17+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in controls | Day 25+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in controls | Day 32+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in controls | Day 39+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in controls | Day 46+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in controls | Day 53+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in controls | Day 60+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 1+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 3+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 5+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 7+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 9+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 11+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 13+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 15+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 17+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 19+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 21+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 23+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 25+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 27+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 29+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 31+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 33+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 35+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 37+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 39+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 41+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 43+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 45+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 47+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 49+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 51+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 53+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 55+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 57+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.
Rate of local and/or systemic occurrence of infection on the PICCline in the experimental group | Day 59+48 hours
  Occurrence of infection on the PICCline, local and/or systemic, and its time of occurrence according to the definition of the Technical Committee on Nosocomial Infections and Healthcare-Associated Infections (CTINILS) during intensive treatment, from the beginning of induction chemotherapy to the beginning of the first consolidation. Local infection will be recorded from the time of PICCline placement, and systemic infection will be recorded when it occurs.

SECONDARY OUTCOMES:
Pain or discomfort generated by PICCline dressing changes in controls | Day 1
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in controls | Day 9
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in controls | Day 17
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in controls | Day 25
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change.
Pain or discomfort generated by PICCline dressing changes in controls | Day 32
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in controls | Day 39
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in controls | Day 46
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in controls | Day 53
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in controls | Day 60
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 1
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 3
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 5
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 7
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 9
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 11
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 13
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 15
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 17
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 19
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 21
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 23
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 25
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 27
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 29
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 31
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 33
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 35
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 37
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 39
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 41
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 43
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 45
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 47
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 49
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 51
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 53
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 55
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 57
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 59
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Pain or discomfort generated by PICCline dressing changes in the experimental group | Day 61
  The patient will be asked to evaluate pain according to a visual analog scale following each dressing change. On this scale, absence of pain = 0 mm and maximum pain imaginable = 100 mm.
Length of time in hospital in controls | At the end of hospitalization
  The duration of time in hospital will be measured from the first day of receiving chemotherapy until transfer towards a healthcare facility for follow-up and rehabilitation or return home.
Length of time in hospital in the experimental group | At the end of hospitalization
  The duration of time in hospital will be measured from the first day of receiving chemotherapy until transfer towards a healthcare facility for follow-up and rehabilitation or return home.
Bacterial species isolated after cytobacteriological analysis of samples (blood cultures and PICCline) and sensitivity to antibiotics in controls | At the end of the 2-month follow-up, on Day 60
  If an infection on the PICCline is suspected, the device will be removed and blood cultures will be taken from the PICCLine and the periphery. If the PICCline culture is positive and the blood cultures negative, the infection is local and device-related. If the PICCline culture and peripheral blood cultures are positive, then catheter-related bacteremia is diagnosed. If general signs like fever appear in a patient with a PICCline without local signs of infection, then blood taken from the periphery and blood from the PICCLine will be cultured. If both blood cultures are positive, catheter-related bacteremia is highly probable. If the blood culture bottle taken from the periphery remains negative and there is a strong suspicion of infection related to the PICCline, then new blood cultures from the periphery and from the device will be performed in order to be able to conclude that there is bacteremia/device colonization/contamination.
Bacterial species isolated after cytobacteriological analysis of samples (blood cultures and PICCline) and sensitivity to antibiotics in the experimental group | At the end of the 2-month follow-up, on Day 60
  If an infection on the PICCline is suspected, the device will be removed and blood cultures will be taken from the PICCLine and the periphery. If the PICCline culture is positive and the blood cultures negative, the infection is local and device-related. If the PICCline culture and peripheral blood cultures are positive, then catheter-related bacteremia is diagnosed. If general signs like fever appear in a patient with a PICCline without local signs of infection, then blood taken from the periphery and blood from the PICCLine will be cultured. If both blood cultures are positive, catheter-related bacteremia is highly probable. If the blood culture bottle taken from the periphery remains negative and there is a strong suspicion of infection related to the PICCline, then new blood cultures from the periphery and from the device will be performed in order to be able to conclude that there is bacteremia/device colonization/contamination.

OTHER OUTCOMES:
Age of patients in the control group | At the inclusion visit (- 48 hours to Day 0)
  In years
Age of patients in the experimental group | At the inclusion visit (- 48 hours to Day 0)
  In years
Body Mass Index of patients in the control group | At the inclusion visit (- 48 hours to Day 0)
  Body Mass Index = Weight ÷ (Height)2
Body Mass Index of patients in the experimental group | At the inclusion visit (- 48 hours to Day 0)
  Body Mass Index = Weight ÷ (Height)2
Patients' medical history : control group | At the inclusion visit (- 48 hours to Day 0)
  The medical history of each patient in the control group will be recorded.
Patients' medical history : experimental group | At the inclusion visit (- 48 hours to Day 0)
  The medical history of each patient in the experimental group will be recorded.
Type of leukemia : control group | At the inclusion visit (- 48 hours to Day 0)
  The type of leukemia of each patient in the control group will be recorded
Type of leukemia : experimental group | At the inclusion visit (- 48 hours to Day 0)
  The type of leukemia of each patient in the experimental group will be recorded
Treatment start date : control group | At the inclusion visit (- 48 hours to Day 0)
  The treatment start date of each patient in the control group will be recorded
Treatment start date : experimental group | At the inclusion visit (- 48 hours to Day 0)
  The treatment start date of each patient in the experimental group will be recorded
Date when patients' aplasia started : control group | At the inclusion visit (- 48 hours to Day 0)
  The date when each patient in the control group started aplasia will be recorded
Date when patients' aplasia started : experimental group | At the inclusion visit (- 48 hours to Day 0)
  The date when each patient in the experimental group started aplasia will be recorded
Date when patients' aplasia ended : control group | End of 2-month follow-up
  The date when each patient in the control group ended their aplasia will be recorded
Date when patients' aplasia ended : experimental group | At the end of the 2-month follow-up, on Day 60
  The date when each patient in the experimental group ended their aplasia will be recorded
Date of hospital discharge : control group | At the end of the 2-month follow-up, on Day 60
  The date when each patient in the control group was discharged from hospital will be recorded.
Date of hospital discharge : experimental group | At the end of the 2-month follow-up, on Day 60
  The date when each patient in the experimental group was discharged from hospital will be recorded.
Antibiotic therapy provided : control group | At the end of the 2-month follow-up, on Day 60
  The antibiotic therapy provided to each patient in the control group will be recorded
Antibiotic therapy provided : experimental group | At the end of the 2-month follow-up, on Day 60
  The antibiotic therapy provided to each patient in the experimental group will be recorded
Presence of parenteral nutrition : control group | At the end of the 2-month follow-up, on Day 60
  For each patient in the control group. Recorded as YES/NO
Presence of parenteral nutrition : experimental group | At the end of the 2-month follow-up, on Day 60
  For each patient in the experimental group. Recorded as YES/NO
Occurrence of thrombosis on the PICCline : control group | At the end of the 2-month follow-up, on Day 60
  For each patient in the control group : YES/NO and date
Occurrence of thrombosis on the PICCline : experimental group | At the end of the 2-month follow-up, on Day 60
  For each patient in the experimental group : YES/NO and date
Device related data : control group | At the end of the 2-month follow-up, on Day 60
  Device-related data: number and types of previous central lines, history of infection, type of device, number of lines, type of fixation, type of dressing, device use protocols, description of puncture site appearance, related intercurrent events, identified germs will be recorded for each patient in the control group.
Device related data : experimental group | At the end of the 2-month follow-up, on Day 60
  Device-related data: number and types of previous central lines, history of infection, type of device, number of lines, type of fixation, type of dressing, device use protocols, description of puncture site appearance, related intercurrent events, identified germs will be recorded for each patient in the experimental group.

CONTACTS AND LOCATIONS:
Overall Officials: Julie LASSALLE, Mme., Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Montpellier Hôpital St-Eloi, Montpellier, France

IPD SHARING:
Plan to Share IPD: No